CLINICAL TRIAL: NCT02429661
Title: Girls First - India Evaluation (2013-2015)
Brief Title: Girls First - India (2013-2015)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CorStone (Other)
Collaborators: David & Lucile Packard Foundation (Unknown); Gramin Evam Nagar Vikas Parishad (GENVP) (Unknown); Integrated Development Foundation Nepal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 01-GF-IN-2013
Record Dates: First submitted 2015-04-22; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Emotional Wellbeing; Social Wellbeing; Physical Wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RC (Girls First Resilience Curriculum) (Experimental): The Girls First Resilience Curriculum is delivered in peer support groups of 12-15 students per group over 23 weekly 1-hour sessions. The curriculum draws from fields such as positive psychology, emotional competence/intelligence, and restorative practices, and aims to improve students' psychosocial assets and wellbeing.
  Interventions: Behavioral: Peer support groups
- HC (Girls First Health Curriculum) (Experimental): The Girls First Health Curriculum is delivered in peer support groups of 12-15 students per group over 21 weekly 1-hour sessions. The curriculum covers topics such as nutrition, sexual and reproductive health, clean water, hygiene, and common diseases, and aims to improve students' physical health and wellbeing.
  Interventions: Behavioral: Peer support groups
- RC+HC (Girls First) (Experimental): Girls First is a combination of the Girls First Resilience Curriculum (RC) and the Girls First Health Curriculum (HC).
  Interventions: Behavioral: Peer support groups
- SC (School-as-usual control) (No Intervention): Participants receive no intervention and attend school as they usually would.

INTERVENTIONS:
Behavioral: Peer support groups
  Arms: HC (Girls First Health Curriculum); RC (Girls First Resilience Curriculum); RC+HC (Girls First)

SUMMARY:
The purpose of this study is to determine the social, emotional, physical, and educational effects of Girls First, a combined resilience and adolescent health program, vs. its components and a control group, among adolescents in India.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at schools or present at sites selected for study
* Must complete consent/assent process

Exclusion Criteria:

* None

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4592 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Psychosocial assets and wellbeing | Change from baseline, measured at program completion (average of 6 months)
  Measured by self-report scales
Physical health and wellbeing | Change from baseline, measured at program completion (average of 6 months)
  Measured by self-report questions

SECONDARY OUTCOMES:
Educational wellbeing | Change from baseline, measured at program completion (average of 6 months)
  Measured by self-report questions

CONTACTS AND LOCATIONS:
Overall Officials: John Peabody, MD, PhD, Principal Investigator — QURE Healthcare
Locations (1):
- CorStone, Mill Valley, California, United States

REFERENCES:
- [Derived] Leventhal KS, DeMaria LM, Gillham J, Andrew G, Peabody JW, Leventhal S. Fostering emotional, social, physical and educational wellbeing in rural India: the methods of a multi-arm randomized controlled trial of Girls First. Trials. 2015 Oct 26;16:481. doi: 10.1186/s13063-015-1008-3. PMID 26503139